CLINICAL TRIAL: NCT06816667
Title: A Phase 1/2 Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate Safety, Tolerability and Efficacy of Multiple Sublingual Microdoses of 5-MeO-DMT in Reducing Symptoms of Depression and/or Anxiety.
Brief Title: Safety, Tolerability, and Efficacy of Sublingual Microdoses of 5-MeO-DMT for Depression and Anxiety
Acronym: 5-MeO-DMT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biomind Labs Inc. (Industry)
Collaborators: Hospital Descentralizado Dr. Marcial V. Quiroga (Unknown); Universidad Católica de Cuyo (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BMND08-01
Record Dates: First submitted 2024-12-10; First posted 2025-02-10 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers
Keywords: 5-MeO-DMT; Sublingual formulation; Safety; Tolerability; Pharmacokinetics; Psychedelics; Double blinded Placebo-controlled; Mood disorders; Phase I/II clinical trial; Efficacy; Anxiety; Depression
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders; Depression | interventions — Methoxydimethyltryptamines; Pharmacokinetics; Vital Signs

STUDY DESIGN:
Intervention Model Description: ThisPhase I/II clinical trial employs a randomized, double-blind, placebo-controlled design to evaluate the safety, pharmacokinetics, and therapeutic potential of sublingual 5-MeO-DMT. Forty healthy volunteers are randomized into four groups: placebo, or 5-MeO-DMT at doses of 6 mg, 9 mg, or 12 mg, receiving weekly doses for four weeks.
  Phase I focuses on safety and pharmacokinetics, monitoring vital signs, ECGs, and biochemical markers while analyzing parameters like Cmax, Tmax, and AUC. Phase II assesses efficacy in reducing anxiety and depression, measured through validated scales (STAI, BDI-II, DASS-21), alongside neurocognitive assessments (FAS, PASAT).
  This trial aims to provide comprehensive data on 5-MeO-DMT's safety, tolerability, and potential therapeutic effects for well being, mood and anxiety disorders.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: 6 mg of 5-MeO-DMT Sublingual Administration (Experimental): In this arm, participants will receive a sublingual dose of 6 mg of 5-MeO-DMT once a week for four consecutive weeks. This dosage is designed to evaluate the safety, tolerability, and potential efficacy of 5-MeO-DMT at a sub-psychedelic level.
  Comprehensive monitoring will include assessments of vital signs, adverse reactions, and overall well-being. Psychiatric evaluations, such as the State-Trait Anxiety Inventory (STAI) and Beck Depression Inventory II (BDI-II), will measure changes in anxiety and depression symptoms. Neurocognitive tests will assess functions like attention, working memory, and executive function.
  EEG evaluations will explore potential changes in brain activity. The findings from this arm will provide critical insights into the effects of a 6 mg dose on emotional health and cognitive performance, contributing to the understanding of 5-MeO-DMT's therapeutic potential in mood and anxiety disorders without inducing a full psychedelic experience.
  Interventions: Drug: BMND08; Procedure: Brain electrical activity monitor; Diagnostic Test: Biochemical determinations; Diagnostic Test: Acute Subjective Ratings of Psychedelic Effects; Diagnostic Test: vital signs; Diagnostic Test: Cognitive Assessments; Diagnostic Test: Psychiatric Assessments
- Arm 2: 9 mg 5-MeO-DMT Sublingual Administration (Experimental): In this arm, participants will receive a sublingual dose of 9 mg of 5-MeO-DMT once a week for four consecutive weeks. This dosage is chosen to evaluate the safety, tolerability, and pharmacokinetics of 5-MeO-DMT at a sub-psychedelic level.
  Participants will be closely monitored for adverse effects, changes in vital signs, and overall health during the treatment period. Assessments will include validated psychiatric evaluations, such as STAI and BDI-II, to measure changes in anxiety and depressive symptoms. Neurocognitive tests, including DSS, FAS and PASAT, will evaluate processing speed and executive function.
  EEG recordings will explore potential changes in brain activity. This arm will provide valuable insights into the emotional and cognitive effects of the 9 mg dose, offering critical information on its therapeutic potential for anxiety and depression while ensuring safety and tolerability without inducing full psychedelic experiences.
  Interventions: Drug: BMND08; Procedure: Brain electrical activity monitor; Diagnostic Test: Biochemical determinations; Diagnostic Test: Acute Subjective Ratings of Psychedelic Effects; Diagnostic Test: vital signs; Diagnostic Test: Cognitive Assessments; Diagnostic Test: Psychiatric Assessments
- Arm 3: 12 mg 5-MeO-DMT Sublingual Administration (Experimental): In this arm, participants will receive a sublingual dose of 12 mg of 5-MeO-DMT once a week for four consecutive weeks. This higher dose is designed to evaluate the safety, tolerability, and pharmacokinetics of 5-MeO-DMT at a level that remains below the threshold for inducing full psychedelic experiences.
  Participants will be closely monitored for adverse effects, changes in vital signs, and overall health during the treatment period. Detailed psychiatric assessments, including the STAI, BDI-II and DASS-21 will be used to measure changes in anxiety, depression, and emotional well-being. Neurocognitive tests, such as the FAS, PASAT and Digit Symbol, to evaluate attention, working memory, and processing speed.
  Additionally, EEG evaluations will explore potential changes in brain activity. Data from this arm will provide critical insights into the therapeutic potential of the 12 mg dose for reducing mood and anxiety symptoms while ensuring safety and maintaining tolerability.
  Interventions: Drug: BMND08; Procedure: Brain electrical activity monitor; Diagnostic Test: Pharmacokinetic Study of Sublingually Administered Psychoactive Substance; Diagnostic Test: Biochemical determinations; Diagnostic Test: Acute Subjective Ratings of Psychedelic Effects; Diagnostic Test: vital signs; Diagnostic Test: Cognitive Assessments; Diagnostic Test: Psychiatric Assessments
- Arm 4: Placebo Sublingual Administration (Placebo Comparator): Participants in this arm will receive a placebo formulation administered sublingually once a week for four consecutive weeks. The placebo is designed to be indistinguishable from the active 5-MeO-DMT formulations in appearance, taste, and administration method, ensuring that both participants and investigators remain blinded to treatment allocations.
  Participants will undergo the same evaluations as those in the active treatment arms. These assessments include psychiatric evaluations (STAI, BDI-II, and DASS-21), and neurocognitive tests to measure attention, memory, and processing speed. EEG evaluations will also be performed to explore potential changes in brain activity.
  This arm serves as the baseline comparator, allowing for the differentiation of the specific therapeutic effects of 5-MeO-DMT from potential placebo effects. The findings will help establish the safety and efficacy of the active compound in reducing symptoms of anxiety and depression.
  Interventions: Drug: BMND08; Procedure: Brain electrical activity monitor; Diagnostic Test: Biochemical determinations; Diagnostic Test: Acute Subjective Ratings of Psychedelic Effects; Diagnostic Test: vital signs; Diagnostic Test: Cognitive Assessments; Diagnostic Test: Psychiatric Assessments

INTERVENTIONS:
Drug: BMND08 — Participants will receive a sublingual dose of 5-MeO-DMT once a week for four consecutive weeks. The intervention will be administered in the form of a sublingual tablet. The substance 5-MeO-DMT, a potent tryptamine, is known for its psychoactive properties but will be administered at a dose that does not induce a full psychedelic experience.
  Other Names: Sublingual Administration of BMND08; 5 MeO-DMT; 5-Methoxy-N,N-dimethyltryptamine
Procedure: Brain electrical activity monitor — EEG is a technique used to monitor brain electrical activity by recording brain waves through electrodes placed on the scalp. This procedure allows the assessment of brain waves such as delta, theta, alpha, and beta, specifically to evaluate the changes in brain activity following sublingual administration of 5-MeO-DMT.
  Other Names: Electroencephalography (EEG)
Diagnostic Test: Pharmacokinetic Study of Sublingually Administered Psychoactive Substance — For pharmacokinetic analysis, approximately 6 mL of EDTA blood will be collected to assess the pharmacokinetics of a sublingual dose of 5-MeO-DMT. Samples will be obtained at baseline (pre-dose, 0 minutes) and at the following time points post-dose: 5, 10, 20, 30, 40, 50, 60, and 120 minutes.
  Other Names: Pharmacokinetics
  Arms: Arm 3: 12 mg 5-MeO-DMT Sublingual Administration
Diagnostic Test: Biochemical determinations — Biochemical determinations will be performed to assess hematological, renal, hepatic, cardiac, and cellular lysis functions. The biochemical markers that will be measured include red blood cells, hematocrit, hemoglobin, glycated hemoglobin, white blood cells, microalbuminuria (urine albumin/creatinine ratio), and various serum markers such as cortisol, glucose, urea, serum creatinine, total cholesterol, HDL, LDL, triglycerides, AST, ALT, lactate dehydrogenase (LDH), creatine kinase (CK), CK-MB, and C-reactive protein.
Diagnostic Test: Acute Subjective Ratings of Psychedelic Effects — To determine the intensity of the acute effects experienced by subjects, retrospective ratings will be collected 1 hour after 5-MeO-DMT or placebo exposure. Subjective ratings will include the Peak Experience Scale (PES), the Ego Dissolution Inventory (EDI), and the Mystical Experiences Questionnaire (MEQ).
Diagnostic Test: vital signs — Vital signs, including blood pressure, heart rate, oxygen saturation, respiration rate, body temperature, and electrocardiograms (ECGs), will be monitored over the six weeks of the treatment
Diagnostic Test: Cognitive Assessments — Cognitive assessments will evaluate the effects of sublingual 5-MeO-DMT on cognitive functions. Participants will undergo the Phonological Verbal Fluency Test (FAS) to assess executive function, the Paced Auditory Serial Addition Test (PASAT) to evaluate processing speed, and the Digit Span Scale (DSS) for attention span and working memory. These tests will be administered at baseline, during treatment, and post-treatment to assess any cognitive changes in response to the different doses of 5-MeO-DMT (6 mg, 9 mg, 12 mg) or placebo, helping to determine how the intervention may influence cognitive processing, memory, and attention.
Diagnostic Test: Psychiatric Assessments — Psychiatric evaluations will be conducted to assess the emotional and psychological effects of sublingual 5-MeO-DMT. Participants will complete the Beck Depression Inventory II (BDI II) to measure mood and depressive symptoms, the State-Trait Anxiety Inventory (STAI) to evaluate state anxiety, and the Depression, Anxiety, and Stress Scale (DASS-21) to assess stress levels. Additionally, the Suicidal Ideation Scale (SSI) will be used to monitor any changes in suicidal ideation throughout the study. These psychiatric assessments will be administered at multiple time points during the study to evaluate the potential therapeutic effects of 5-MeO-DMT in improving mood, anxiety, and overall psychological well-being.

SUMMARY:
This Phase I/II clinical trial investigates the safety, tolerability, and potential therapeutic benefits of a novel sublingual formulation of 5-MeO-DMT. The study uses a randomized, double-blind, placebo-controlled design to evaluate the compound's effects on mood and overall well-being, focusing on participants with elevated symptoms of anxiety and depression.

Study Design and Objectives:

Participants are divided into four groups: one receiving a placebo and three receiving different doses of 5-MeO-DMT (6 mg, 9 mg, or 12 mg). Each group comprises 10 participants, totaling 40 individuals. The study administers one dose weekly for four weeks, with comprehensive monitoring at baseline and throughout the trial to track changes in emotional, cognitive, and physical well-being.

Objectives:

Assessing 5-MeO-DMT's impact on anxiety, depression, and emotional well-being. Understanding its pharmacokinetics (absorption, distribution, metabolism, and excretion).

Evaluating its safety profile and identifying potential side effects, both mild and severe.

Monitoring and Safety Participant safety is prioritized, with medical professionals conducting regular evaluations of vital signs, such as heart rate and blood pressure. Detailed tracking of mood, perception, and physical responses ensures any adverse reactions are documented and analyzed.

Sublingual Administration The sublingual route is being studied for its rapid absorption into the bloodstream. Researchers will determine how efficiently the body processes 5-MeO-DMT, its duration in the bloodstream, and its influence on daily life. These findings will inform the practicality of this administration method in clinical settings.

Significance of the Study This trial aims to establish a robust safety and tolerability profile for 5-MeO-DMT while exploring its effects on anxiety and depression. The results will also provide essential data to guide future studies into its therapeutic potential for improving mental health and overall quality of life.

By addressing both the compound's safety and potential benefits, this research lays the groundwork for developing innovative mental health treatments.

DETAILED DESCRIPTION:
This Phase I/II clinical trial employs a rigorous, randomized, double-blind, placebo-controlled design to evaluate the safety, tolerability, pharmacokinetics, and efficacy of a novel sublingual formulation of 5-MeO-DMT. The trial focuses on understanding the compound's effects in healthy volunteers and those with elevated symptoms of anxiety and depression, aiming to build a comprehensive profile of its potential therapeutic and pharmacological properties.

Study Objectives

The Phase I component emphasizes:

* Safety and Tolerability: Assessing physiological responses, including vital signs (heart rate, blood pressure, respiration rate, temperature) and cardiac function (ECGs). Biochemical markers of renal, hepatic, and hematological health will be monitored to detect potential adverse effects.
* Pharmacokinetics: Evaluating how 5-MeO-DMT is absorbed, distributed, metabolized, and eliminated through blood sampling at multiple time points. Key metrics include peak plasma concentration (Cmax), time to peak (Tmax), and overall exposure (AUC).

The Phase II component explores the efficacy of 5-MeO-DMT in reducing symptoms of anxiety and depression and enhancing emotional well-being.

Participants and Dosing Regimen The trial enrolls 40 participants aged 40-80, divided into four groups: one placebo group and three active treatment groups receiving sublingual doses of 6 mg, 9 mg, or 12 mg of 5-MeO-DMT. A single weekly dose is administered over four weeks, enabling the evaluation of immediate and cumulative effects.

Recruitment will target healthy volunteers who meet specific anxiety and mood criteria. Notably, participants will be screened to exclude individuals with previous psychedelic experiences involving tryptamines, ergolines, or phenethylamines, those with contraindications to the use of psychedelics, and those currently taking prescribed psychoactive medications. This includes serotonin reuptake inhibitors, benzodiazepines, medications primarily affecting serotonin neurons (e.g., ondansetron), and MAO inhibitors.

Neurocognitive and Psychological Assessments

Participants undergo validated assessments to evaluate changes in:

* Mood and Anxiety: Tools include the State-Trait Anxiety Inventory (STAI), Beck Depression Inventory II (BDI-II), Depression, Anxiety, and Stress Scale (DASS-21), and Suicidal Ideation Scale (SSI).
* Cognitive Function: Neurocognitive tests like the Phonological Verbal Fluency Test (FAS), Paced Auditory Serial Addition Test (PASAT), and Digit Span Scale (DSS) assess executive function, working memory, and attention.

Validated instruments will be employed to evaluate mood, anxiety levels, cognitive function, and any perceptual or psychological effects experienced by participants. These assessments will be conducted at baseline (Week 0), during each dosing week (Weeks 1-4), and at the end of the study (Week 5). By measuring these parameters, the trial aims to identify the effects of sub-psychedelic doses of 5-MeO-DMT on cognitive processes and emotional states.

Safety Protocols The study complies with Good Clinical Practice (GCP) and ethical standards, including approval from the CEI of the Ministry of Health of San Juan, Argentina. Informed consent is obtained from all participants, who are screened to exclude individuals with prior psychedelic experiences, contraindications, or concurrent use of psychoactive medications.

The trial prioritizes participant safety with continuous monitoring and immediate medical response protocols for any adverse events.

Expected Outcomes This study aims to generate a comprehensive dataset on the safety, pharmacokinetics, and potential efficacy of sublingual 5-MeO-DMT, providing a clear and detailed understanding of its safety and tolerability profile under controlled conditions.

The findings are expected to inform future research into the therapeutic potential of 5-MeO-DMT for anxiety, depression, and other mental health disorders, offering critical insights into its clinical applications. By advancing the understanding of psychedelic compounds, this study represents a pivotal step toward developing innovative, evidence-based treatments for mental health challenges.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participants aged between 40 and 80 years, regardless of sex.
* Must provide written informed consent to participate in the study.
* Participants must exhibit moderate to high levels of anxiety and/or depression:
* Anxiety levels assessed using the State-Trait Anxiety Inventory (STAI):
* STAI-S (State) score of ≥20 for men and ≥23 for women
* STAI-T (Trait) score of ≥20 for men and ≥26 for women
* Depression levels assessed using the Beck Depression Inventory (BDI):
* BDI score of ≥21 indicating the presence of moderate to severe depressive symptoms.
* Participants may meet the criteria for either anxiety, depression, or both, as long as they meet the respective thresholds for each

Exclusion Criteria:

* Liver dysfunction
* Cardiovascular conditions, including: Uncontrolled hypertension, Angina, Clinically significant ECG abnormalities (e.g., atrial fibrillation), Transient ischemic attack (TIA) within the last 6 months.
* Stroke or peripheral/pulmonary vascular disease without active claudication.
* Blood pressure exceeding 140 mmHg systolic or 90 mmHg diastolic.
* Epilepsy or a history of seizures.
* Kidney failure.
* Insulin-dependent diabetes.
* Chronic obstructive pulmonary disease (COPD).
* Increased intracranial or cerebrospinal pressure
* Hyperthyroidism
* Psychotic symptoms or a family history of psychotic disorders
* Prodromal symptoms of schizophrenia or dissociative identity disorder.
* Severe symptoms of depression or anxiety requiring immediate treatment with antidepressants or daily anxiolytic medications, especially in cases involving suicidal ideation.
* Medications: Regular use of prescribed psychoactive medications, such as: Benzodiazepines, Medications affecting serotonin neurons (e.g., ondansetron), Monoamine oxidase inhibitors (MAOIs).
* Drug Interactions: Use of potent metabolic inducers or inhibitors, including: Inducers: Rifampicin (rifabutin, rifapentine), anticonvulsants (carbamazepine, phenytoin, phenobarbital), nevirapine, efavirenz, taxol, dexamethasone. or Inhibitors: All HIV protease inhibitors, itraconazole, ketoconazole, erythromycin, clarithromycin, and troleandomycin.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events Coded by MedDRA Following Sublingual Administration of 5-MeO-DMT | Throughout the 6 weeks of the interventional study.
  Number of participants experiencing Adverse Events following the sublingual administration of 5-MeO-DMT, as assessed and coded by MedDRA.
Maximum Plasma Concentration (Cmax) following sublingual administration of 5-MeO-DMT. | From baseline at 0 minutes to 120 minutes following administration.
  Blood samples will be collected prior to and up to 120 minutes post-administration to determine the peak plasma concentration (Cmax) of 5-MeO-DMT.
Time to Maximum Plasma Concentration (Tmax) following sublingual administration of 5-MeO-DMT | From baseline at 0 minutes to 120 minutes following administration.
  Blood samples will be collected to assess the time taken to reach the maximum plasma concentration (Tmax) of 5-MeO-DMT.
Area Under the Curve (AUC) following sublingual administration of 5-MeO-DMT. | From baseline at 0 minutes to 120 minutes following administration.
  Blood samples will be analyzed to calculate the area under the plasma concentration-time curve (AUC), reflecting the overall drug exposure.
Elimination Half-life (t1/2) of 5-MeO-DMT. | From baseline at 0 minutes to 120 minutes following administration.
  Blood samples will be used to determine the elimination half-life (t1/2) of 5-MeO-DMT after sublingual administration.
Mystical Experience Questionnaire (MEQ) Assessment at 40 Minutes Post-Administration | The MEQ will be completed at 40 minutes post-administration during each dosing week (Weeks 1-4) to assess the subjective mystical experiences induced by sublingual 5-MeO-DMT.
  The Mystical Experience Questionnaire (MEQ) is used to assess the subjective mystical experiences following psychedelic administration. It evaluates aspects such as feelings of unity, transcendence, and the sense of the sacred. The MEQ includes questions about altered perceptions of time, space, and self, as well as emotional and cognitive shifts. Higher scores indicate a stronger experience of mystical qualities.
Peak Experience Scale (PES) Assessment at 40 Minutes Post-Administration | The PES will be completed at 40 minutes post-administration during each dosing week (Weeks 1-4) to capture the intensity and emotional impact of the 5-MeO-DMT experience.
  The Peak Experience Scale (PES) is a tool for measuring the intensity and quality of peak experiences following psychedelic use. It includes items related to emotional intensity, personal insight, and transcendence. Participants rate the emotional and psychological impact of their experiences, with higher scores reflecting more intense peak experiences.
Ego Dissolution Inventory (EDI) Assessment at 40 Minutes Post-Administration | The EDI will be completed at 40 minutes post-administration during each dosing week (Weeks 1-4) to evaluate the degree of ego dissolution experienced after 5-MeO-DMT consumption.
  The Ego Dissolution Inventory (EDI) assesses the extent to which participants experience a loss of ego boundaries or self-identity following psychedelic administration. It includes questions that explore the feeling of oneness with the environment, other people, or the universe, as well as the dissolution of self-related thoughts and ego. Higher scores indicate stronger experiences of ego dissolution.

SECONDARY OUTCOMES:
Mean change in Beck Depression Inventory II (BDI-II) from Baseline to Week 5 | The BDI test will be conducted at baseline (Week 0), during treatment (Weeks 1-4), and at follow-up (Week 5) to assess the impact of 5-MeO-DMT on the severity of depression.
  The Beck Depression Inventory II (BDI-II) is a 21-item self-report questionnaire designed to assess the severity of depressive symptoms. Each item is scored from 0 to 3, with the total score ranging from 0 to 63. Higher scores indicate more severe depression.
Mean change in State-Trait Anxiety Inventory (STAI) from Baseline to Week 5 | STAI evaluations will be conducted at baseline (Week 0), during treatment (Weeks 1-4), and at follow-up (Week 5) to assess the impact of 5-MeO-DMT on anxiety levels.
  The State-Trait Anxiety Inventory (STAI) is a 40-item scale that measures both state anxiety (current feelings of anxiety) and trait anxiety (general tendency to experience anxiety). Each item is scored from 1 to 4, with the overall score ranging from 20 to 80. Higher scores indicate higher levels of anxiety.
Mean change in Depression, Anxiety, and Stress Scale (DASS-21) from Baseline to Week 5 | DASS-21 will be conducted at baseline (Week 0), during treatment (Weeks 1-4), and at follow-up (Week 5) to evaluate the impact of 5-MeO-DMT on mood and stress.
  The Depression, Anxiety, and Stress Scale (DASS-21) is a 21-item questionnaire that measures the severity of depression, anxiety, and stress symptoms. Each item is scored from 0 to 3, with higher scores indicating more severe symptoms. The total score ranges from 0 to 63.
Change in Phonological Verbal Fluency Test (FAS) from Baseline to Week 5 | The FAS will be administered at baseline (Week 0), during treatment (Weeks 1-4), and at follow-up (Week 5) to assess changes in executive function during and after sublingual 5-MeO-DMT administration.
  The Phonological Verbal Fluency Test (FAS) measures executive function by assessing a participant's ability to generate words within a specific time limit, categorized by a starting letter. The task is designed to evaluate verbal memory, cognitive flexibility, and processing speed. The FAS ranges from 0 to the maximum number of words generated in 1 minute. A higher score indicates better performance.
Change in Paced Auditory Serial Addition Test (PASAT) from Baseline to Week 5 | The PASAT will be administered at baseline (Week 0), during treatment (Weeks 1-4), and at follow-up (Week 5) to evaluate the effects of 5-MeO-DMT on cognitive processing speed and attention.
  The Paced Auditory Serial Addition Test (PASAT) is a cognitive test used to measure processing speed and attention. Participants are presented with a sequence of 60 numbers, each separated by 2 seconds, and must add each new number to the previous one as quickly as possible. Performance is scored based on the percentage of correct responses within the given time. The PASAT ranges from 0 to 100. A higher score reflects better cognitive processing and attention.
Change in Digit Span Scale (DSS) from Baseline to Week 5 | The DSS will be administered at baseline (Week 0), during treatment (Weeks 1-4), and at follow-up (Week 5) to assess changes in attention and working memory following 5-MeO-DMT administration.
  The Digit Span Scale (DSS) is used to assess attention span and working memory. In this test, participants must repeat a series of numbers either in the same order (forward) or in reverse (backward). The DSS measures short-term memory and cognitive flexibility. The DSS ranges from 0 to 48. A higher score indicates better working memory and attention capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Martin A. Bruno, PhD, Principal Investigator — Biomind Labs Inc.
Locations (1):
- Hospital Descentralizado Dr. Marcial V. Quiroga., San Juan, Rivadavia, Argentina

IPD SHARING:
Plan to Share IPD: Yes
The study is committed to enhancing scientific research by planning to share individual participant data, aiming to contribute valuable insights to the research community. We will provide a detailed data dictionary alongside the IPD, outlining the variables and types of data collected for each participant, facilitating comprehensive analysis by researchers.
  Specifically, we plan to share all IPD collected throughout the trial, including data that underlie published results. Importantly, all personal information and identifying details of participants will remain strictly confidential and will not be disclosed. This commitment ensures the privacy of individuals involved while still enabling meaningful contributions to scientific knowledge.
  If a decision regarding data sharing is not yet finalized, we will communicate this clearly along with the reasons. Through this approach, we aim to promote transparency in research while maintaining the highest ethical standards for participant data.
Supporting Information: Study Protocol, ICF
Time Frame: The individual participant data (IPD) and any supporting information will be made available starting 6 months after the publication of the study results. This will allow sufficient time for data analysis and the dissemination of primary findings. The data will remain available for at least 5 years following the publication, ensuring ample time for other researchers to access and utilize the data for further analysis or related studies. In case of any modifications to the availability period, these will be communicated clearly along with the reasons. This time frame is subject to ethical and regulatory requirements and may be adjusted if necessary.
Access Criteria: Researchers seeking access to the individual participant data (IPD) and supporting information must submit a formal request outlining their proposed analyses. This proposal should detail the types of analyses, including the statistical methods to be used, which will be reviewed for scientific merit and methodological rigor. A signed data sharing agreement will be required, and the request must be submitted through the designated data sharing platform or by email to the study's data management team. Access to IPD will be granted based on ethical review and approval, ensuring that the proposed research aligns with the study's objectives and respects participant confidentiality. All requests will be reviewed by an independent committee responsible for overseeing data sharing, ensuring transparency, and safeguarding participant privacy.

REFERENCES:
- [Derived] Bistue Millon MB, Noguera L, Bruno D, Vita L, Zanino M, Kassuha DE, Ortiz JE, Feresin GE, Diaz-Dellavalle P, Orosco L, Garces MA, Diez P, Albarracin SG, Bruno MA. Safety and tolerability of multiple sublingual microdoses of 5-MeO-DMT in adults with moderate symptoms of depression and/or anxiety: a randomized, double-blind, placebo-controlled study. Neuropsychopharmacology. 2025 Oct;50(11):1715-1723. doi: 10.1038/s41386-025-02167-3. Epub 2025 Jul 15. PMID 40659913
- See also: Biomind Labs is developing the next generation of pharmaceuticals to treat patients suffering from neurological disorders. This unique approach targets the original and initial drivers of the diseases. — https://www.biomindlabs.com/